CLINICAL TRIAL: NCT01287091
Title: An Open-Label, 3-Part Study to Determine the Relative Bioavailability of Capsule and Tablet Formulations of GDC-0980, the Effect of Food, and the Effect of Rabeprazole on the Pharmacokinetics of the Tablet
Brief Title: A 3-Part Study to Determine the Relative Bioavailability of Capsule and Tablet Formulations of GDC-0980, the Effect of Food, and the Effect of Rabeprazole on the Pharmacokinetics of the Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIM4930g
Record Dates: First submitted 2011-01-07; First posted 2011-02-01 (Estimated); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — 1-(4-((2-(2-aminopyrimidin-5-yl)-7-methyl-4-morpholinothieno(3,2-d)pyrimidin-6-yl)methyl)piperazin-1-yl)-2-hydroxypropan-1-one; Rabeprazole

ARMS (4):
- Part 1 (Experimental)
  Interventions: Drug: GDC-0980
- Part 2 (Experimental)
  Interventions: Drug: GDC-0980
- Part 3: Group A (Experimental)
  Interventions: Drug: GDC-0980; Drug: rabeprazole
- Part 3: Group B (Experimental)
  Interventions: Drug: GDC-0980; Drug: rabeprazole

INTERVENTIONS:
Drug: GDC-0980 — Oral tablet dose
  Arms: Part 1
Drug: GDC-0980 — Oral capsule dose
  Arms: Part 1
Drug: GDC-0980 — Oral tablet dose in fed state
  Arms: Part 2
Drug: GDC-0980 — Oral repeating dose in fasting state
  Arms: Part 3: Group A
Drug: GDC-0980 — Oral repeating dose in fed state
  Arms: Part 3: Group B
Drug: GDC-0980 — Oral tablet in a fasting state
  Arms: Part 2
Drug: rabeprazole — Oral repeating dose
  Arms: Part 3: Group A; Part 3: Group B

SUMMARY:
This will be a single-center, open-label, 3 part study. The study is designed to determine the relative bioavailability of GDC-0980 capsule and tablet formulations under fasting conditions, the effects of a high-fat (fed) meal on the pharmacokinetics of the GDC-0980 tablet, and the effects of rabeprazole on the pharmacokinetics of the GDC-0980 tablet in the presence or absence of a high-fat meal.

ELIGIBILITY:
Inclusion Criteria

* Nonsmoking with a body mass index of 18 to 32 kg/m2
* Medically healthy as determined by the absence of clinically significant findings in the physical examination, medical history, vital sign measurements, clinical laboratory tests, or 12-lead electrocardiograms (ECGs)
* Nonchildbearing potential, defined as either postmenopausal and without recent history of menorrhea or surgically sterile

Exclusion Criteria

* History or clinical manifestations of significant metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, endocrine, gastrointestinal, urological, neurological, or psychiatric disorders, or cancer
* History of inflammatory arthritis
* History of symptomatic hypotension
* History of severe physical injury, direct impact trauma, or neurological trauma within 6 months prior to study start
* History of seizure disorders
* History of bipolar or major depressive disorder
* History of stomach or intestinal surgery or resection that could potentially alter absorption and/or excretion of orally administered drugs with the exception of appendectomy, hernia repair, and cholecystectomy, which are allowed
* History or presence of an abnormal ECG
* History of ventricular dysrhythmias or risk factors for ventricular dysrhythmias
* Abnormality on the chest x-ray at Screening
* History of alcoholism, drug abuse, or drug addiction
* Used any nicotine-containing or nicotine-replacement products within 6 months prior to study start
* Participated in any other investigational drug study in which receipt of an investigational study drug occurred within 1 month or 5 half-lives prior to study start
* Used any prescription medications/products including monoamine oxidase inhibitors, thioridazine, pimozide, or antidepressants within 1 month (2 weeks for antibiotics) prior to study start, with the exception of hormone-replacement therapy or 2 weeks' use of narcotics for pain
* Received any vaccination or immunization within 1 month prior to study start
* Used PPIs or histamine H2-receptor antagonists within 1 month prior to study start
* Hypersensitivity to rabeprazole, or any of its components, or to derived products of benzimidazoles (for Part 3 only)
* Poor peripheral venous access
* Received blood products within 2 months prior to study start
* Positive urine drug or alcohol screen
* Positive screen for hepatitis B surface antigen, hepatitis C virus, or human immunodeficiency virus types 1 and 2
* Unable to consume a high-fat meal (for Parts 2 and 3 only)
* Acute or chronic condition that would limit the subject's ability to complete or participate in this clinical study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-10-14 (Actual); Primary Completion 2011-02-03 (Actual); Study Completion 2011-02-03 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration | Up to day 10
Time to maximum observed plasma concentration | Up to day 10
Plasma half-life | Up to day 10
Oral clearance | Up to day 10
Volume of distribution | Up to day 10
Minimum plasma concentration | Up to day 10

SECONDARY OUTCOMES:
Incidence of adverse events | Up to day 68
Nature of adverse events | Up to day 68
Severity of adverse events | Up to day 68

CONTACTS AND LOCATIONS:
Overall Officials: Scott Holden, M.D., Study Director — Genentech, Inc.
Locations (1):
- Investigational Site, Austin, Texas, United States